CLINICAL TRIAL: NCT01117285
Title: Implementation and Evaluation of an Effective Community Occupational Therapy in Dementia (COTiD) Program
Brief Title: Implementation and Evaluation of the COTiD Program in the Netherlands
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Collaborators: HAN University of Applied Sciences (Other)
Responsible Party: Dr. M.J.L. Graff / Senior research fellow, lecturer, Scientific Institute for Quality of Healthcare (IQ healthcare), Radboud University Nijmegen Medical Centre
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 80-82315-98-090010
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-03

CONDITIONS: Dementia
Keywords: Occupational Therapy; Evidence-Based Practice; Continuing Education; utilization; Guideline; Dementia; Guideline implementation
MeSH Terms: conditions — Dementia; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3-day post-graduate course (Active Comparator): 3-day post-graduate course on the use of the COTiD program in clinical practice
  Interventions: Other: 3-day post-graduate course
- Combined implementation strategy (Experimental): The combined implementation strategy
  Interventions: Other: Combined implementation strategy

INTERVENTIONS:
Other: 3-day post-graduate course — A 3-day course in using the COTiD program in clinical practice. The 3 days are not provided uninterrupted but there are at least two weeks between each day to provide time to practice with the guideline (for discussion on the 2nd day).
  The course consists of theory on the content of the guideline and its effectiveness, Practice parts of the guideline by rol playing, and discussing each others skills through watching video material.
  Other Names: educational strategy
  Arms: 3-day post-graduate course
Other: Combined implementation strategy — The combined implementation strategy provides strategies for occupational therapists (OTs), physicians, and managers.
  OTs receive:
  * 3-day post-graduate course
  * 2 extra training days: Lectures and skills practice focused on using the COTiD program and promoting the use of the program within their organization and network.
  * Coaching on the job: Barriers to using the COTiD program in practice are discussed using motivational interviewing.
  * Discussion platform
  * Web-based registration system: Provides guidance in using the COTiD program for every individual client.
  * Regional meetings: successes and difficulties in using the COTiD are discussed.
  Managers and physicians receive:
  * Information on the COTiD program through a website and newsletters.
  * Motivational reminders.
  Other Names: implementation training
  Arms: Combined implementation strategy

SUMMARY:
The main purpose of this cluster randomized controlled trial is to evaluate the difference in effectiveness between a combined implementation strategy and an educational strategy on the implementation of a community occupational therapy program for clients with dementia and their primary caregivers.

DETAILED DESCRIPTION:
Dementia is associated with a major decrease in quality of life of clients and their caregivers and a major driver of costs in health care. Recently, evidence was found for the effectiveness and cost-effectiveness of a community-based occupational therapy (OT) intervention for older adults with dementia and their caregivers (COTiD program). This intervention resulted in significant improvements in both clients' and caregivers' daily functioning, quality of life, mood and health status. In addition, caregivers experienced an increased sense of competence.

Currently occupational therapists (OTs) are trained in using the program during a 3-day course. In a pilot implementation study it was found that this course was not effective enough as only 20% of the OTs actually used the COTiD program in practice because of a lack of implementation skills, feedback and organisational barriers. In order to increase the use of this program and increase the quality of care a new implementation strategy is developed. This combined implementation strategy provides the OTs with two implementation training days, coaching on the job, regional meetings, discussion platform, web-based registration system and newsletters. In addition physicians and managers are provided with extra information on the COTiD program.

The current study is designed primarily to evaluate the following research questions:

* What is the difference in adherence to the community OT guideline in dementia between OTs receiving the combined implementation strategy and OTs receiving the educational strategy?
* What is the difference in community OT use(referral rate + actual provision of OT) between clusters provided with the combined implementation strategy and clusters provided with the educational strategy?
* What is the difference in cost-effectiveness between the combined implementation strategy and the educational strategy with regard to adherence of OTs to the community OT guideline?

In addition the effect of the implementation strategies on patient and caregiver outcomes will also be measured.

ELIGIBILITY:
Because of the clustered design, there are inclusion and exclusion criteria for clusters as well as for clients with dementia and their caregivers.A cluster is a unit that exists of at least one occupational therapist, one physician, and one manager.

Criteria for clusters

Inclusion Criteria:

* The organization provides outpatient OT.
* The organization expects that they will be able to include a minimum of 8 clients in the study.
* There are at least two OTs, one manager, and one physician willing and able to participate in the study.

Exclusion Criteria:

* The organization does not provide OT or outpatient treatment and is not allowed to refer to OT services in their area that do provide community OT.
* Less than 8 clients are available per year to refer to the OT.
* Physicians, managers or OTs are not willing to participate
* Members of the board of directors responsible for the organization do not agree to participate

Criteria for client with dementia and their informal caregiver

Inclusion Criteria for clients and informal caregivers:

* Client has mild to moderate dementia (MMSE score 10-24, DSM IV criteria for dementia)
* Client lives at home
* Client has an informal caregiver who takes care of the client at least twice a week

Exclusion criteria for clients:

* Client is in a severe stage of dementia
* Client has a depression (GDS (version 30) >12)
* Client has severe behavioral or psychological symptoms in dementia (BPSD)
* Client has a severe illness at the time of inclusion

Exclusion criteria for informal caregivers:

* The caregiver is not able to participate in the OT treatment (e.g. due to illness).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Adherence of occupational therapists to the COTiD program | one year (baseline, T1, and T2)
  Adherence is measured using vignettes. Vignettes are realistic case descriptions about which occupational therapists are asked to answer open ended questions.
Community occupational therapy use according to the COTiD program | one year
  Community OT use reflects:
  * How many people with dementia were referred to OT services in total
  * How many people with dementia were referred specifically to OT according to the COTiD program.
Costs of the implementation strategies | October 2009 - December 2011
  The following cost data is collected:
  Costs of the implementation strategies
  * Costs made by the OTs, managers, and physicians receiving the combined implementation strategy.
  * Costs made by the OTs receiving only the educational strategy.
  * Development and execution costs of the combined implementation strategy.
  * development and execution costs of the educational strategy.
  Costs made buy the cliënt and caregiver
  * Costs made by client and caregiver (using the RUD Lite instrument)regarding healthcare consumption
  * Time the caregiver spends om informal care

SECONDARY OUTCOMES:
Knowledge of the healthcare professionals about the COTiD program | one year (baseline, T1, and T2)
  measured using a multiple choice knowledge test on the most important aspects of the COTiD program.
COTiD program treatment outcome on client and caregiver level | one year (baseline, T1, and T2)
  The following outcomes are evaluated:
  * Clients'processing skills (Assessment of Motor and Process Skills)
  * Need for assistance in daily activities (Interview of Deterioration of Daily Activities in Dementia)
  * Caregivers Sense of Competence (Sense of Competense Questionnaire)
  * Client and caregiver quality of life (EQ5D and Dementia Quality of Life Scale)
  * Client and caregiver self-perceived performance and satisfaction (Canadian Occupational Performance Measure)

CONTACTS AND LOCATIONS:
Overall Officials: Myrra Vernooij-Dassen, PhD, Study Chair — Radboud University Medical Center; Maud Graff, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Scientific Institute for Quality of Healthcare (IQ healthcare) (and 45 Dutch organisation), Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Graff MJ, Vernooij-Dassen MJ, Thijssen M, Dekker J, Hoefnagels WH, Rikkert MG. Community based occupational therapy for patients with dementia and their care givers: randomised controlled trial. BMJ. 2006 Dec 9;333(7580):1196. doi: 10.1136/bmj.39001.688843.BE. Epub 2006 Nov 17. PMID 17114212
- [Background] Graff MJ, Adang EM, Vernooij-Dassen MJ, Dekker J, Jonsson L, Thijssen M, Hoefnagels WH, Rikkert MG. Community occupational therapy for older patients with dementia and their care givers: cost effectiveness study. BMJ. 2008 Jan 19;336(7636):134-8. doi: 10.1136/bmj.39408.481898.BE. Epub 2008 Jan 2. PMID 18171718
- [Background] Voigt-Radloff S, Graff M, Leonhart R, Schornstein K, Vernooij-Dassen M, Olde-Rikkert M, Huell M. WHEDA study: effectiveness of occupational therapy at home for older people with dementia and their caregivers--the design of a pragmatic randomised controlled trial evaluating a Dutch programme in seven German centres. BMC Geriatr. 2009 Oct 2;9:44. doi: 10.1186/1471-2318-9-44. PMID 19799779
- [Background] Graff MJ, Vernooij-Dassen MJ, Thijssen M, Dekker J, Hoefnagels WH, Olderikkert MG. Effects of community occupational therapy on quality of life, mood, and health status in dementia patients and their caregivers: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2007 Sep;62(9):1002-9. doi: 10.1093/gerona/62.9.1002. PMID 17895439
- [Derived] Dopp CM, Graff MJ, Teerenstra S, Olde Rikkert MG, Nijhuis-van der Sanden MW, Vernooij-Dassen MJ. Effectiveness of a training package for implementing a community-based occupational therapy program in dementia: a cluster randomized controlled trial. Clin Rehabil. 2015 Oct;29(10):974-86. doi: 10.1177/0269215514564699. Epub 2014 Dec 28. PMID 25547113
- [Derived] Dopp CM, Graff MJ, Teerenstra S, Nijhuis-van der Sanden MW, Olde Rikkert MG, Vernooij-Dassen MJ. Effectiveness of a multifaceted implementation strategy on physicians' referral behavior to an evidence-based psychosocial intervention in dementia: a cluster randomized controlled trial. BMC Fam Pract. 2013 May 30;14:70. doi: 10.1186/1471-2296-14-70. PMID 23718565
- [Derived] Dopp CM, Graff MJ, Teerenstra S, Adang E, Nijhuis-van der Sanden RW, Olderikkert MG, Vernooij-Dassen MJ. A new combined strategy to implement a community occupational therapy intervention: designing a cluster randomized controlled trial. BMC Geriatr. 2011 Mar 30;11:13. doi: 10.1186/1471-2318-11-13. PMID 21450063